CLINICAL TRIAL: NCT07240233
Title: Implementation of Musical Intervention as a Non-Pharmacological Strategy for Mitigating Anxiety in Dental Procedures
Brief Title: Musical Intervention for Dental Anxiety
Acronym: MI-DENT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Egas Moniz - Cooperativa de Ensino Superior, CRL (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NP110925
Record Dates: First submitted 2025-10-02; First posted 2025-11-20 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Dental Anxiety
Keywords: Dental anxiety; Dental fear; Odontophobia; Music therapy; Therapeutic music listening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music via headphones (Experimental): Participants wear wireless, supra-aural headphones delivering a standardized playlist of classical and baroque pieces
  Interventions: Other: Music via headphones
- Headphones without audio (Active Comparator): Participants wear the same model headphones with no audio to provide passive attenuation of ambient noise
  Interventions: Other: Headphones without audio
- Standard care (No Intervention): no headphones or music; routine dental care proceeds per usual practice

INTERVENTIONS:
Other: Music via headphones — Wear wireless, supra-aural headphones delivering a standardized playlist of classical and baroque pieces
  Arms: Music via headphones
Other: Headphones without audio — wear the same model headphones with no audio to provide passive attenuation of ambient noise
  Arms: Headphones without audio

SUMMARY:
The goal of this clinical trial is to learn if listening to music during dental procedures lowers anxiety in adults. The main questions it aims to answer are: does music during the procedure lower dental anxiety, and does wearing headphones without audio to reduce ambient noise also lower dental anxiety. Researchers will compare three groups to see these effects: music via headphones, headphones without audio, and standard care without headphones or music.

Participants will:

* Complete a short anxiety questionnaire before the dental procedure.
* Receive one of the three approaches during the procedure: music via headphones, headphones without audio, or no headphones/music.
* Complete a short anxiety questionnaire after the dental procedure.

DETAILED DESCRIPTION:
Design and setting This study is a randomized, parallel-group clinical trial conducted in a dental clinic setting, evaluating two non-pharmacological auditory strategies versus standard care for reducing state anxiety during routine dental procedures in adults. Participants are randomized in a 1:1:1 ratio to: music via headphones during the procedure; headphones worn without audio to attenuate ambient noise; or standard care with no headphones or music. State anxiety is measured immediately before and after the clinical encounter to estimate within-person change and between-group differences

Participants Adults receiving dental care at a university-affiliated clinic are approached at chairside prior to seating for eligibility screening and consent. Inclusion criteria include legal age and ability to complete self-report measures independently; key exclusions include hearing impairment or hearing aids, sedative medication use prior to the visit, cognitive impairment limiting informed consent, or refusal to consent. Recruitment occurs consecutively during routine clinical sessions to enhance generalizability to real-world practice.

Interventions

* Music via headphones: participants wear wireless, supra-aural headphones delivering a standardized playlist of classical and baroque pieces (fixed sequence, ~3-hour list; actual exposure limited to visit length). Communication needs are accommodated by temporarily removing headphones when signaled; patients are instructed to raise the left hand to request interaction or report discomfort; headphones may be removed for imaging or clinical needs.
* Headphones without audio: participants wear the same model headphones with no audio to provide passive attenuation of ambient noise; clinical communication procedures mirror the music arm.
* Standard care: no headphones or music; routine dental care proceeds per usual practice.

Equipment and hygiene Wireless supra-aural Bluetooth 5.0 headphones with padded cushions are used to maximize comfort and passive noise isolation and to avoid cable interference with dental equipment. After each session, headphones are disinfected using 70% isopropyl alcohol wipes on all skin-contact surfaces and allowed to dry before reuse, following basic device-compatible infection control practices.

Outcomes and timing State dental anxiety and general state anxiety are assessed immediately pre-procedure and post-procedure using validated self-report instruments routinely used in dental anxiety research; higher scores indicate greater anxiety, and change scores (post minus pre) are the primary comparisons across arms. Pre-procedure sociodemographic and screening items characterize the sample and capture potential confounders (for example, psychotropic use, prior psychiatric diagnosis, prior anxiety crises in dental settings).

Randomization and masking Allocation to the three arms uses simple random assignment at participant level prior to the start of the procedure; outcome assessors use standardized, self-administered questionnaires to minimize assessor influence, but masking of participants and providers is not feasible due to the nature of the interventions. Analyses will follow the intention-to-treat principle, with sensitivity analyses as needed for protocol deviations.

Data handling and analysis Data are captured into a secured database for statistical analysis using standard software; descriptive statistics summarize the sample and visit characteristics (for example, procedure type and duration). The main analysis compares anxiety change across arms using repeated-measures multivariate methods to test group, time, and group-by-time interaction effects, which can increase power by accounting for within-person correlation and simultaneous outcomes when applicable. Planned covariates include procedure category (for example, emergency care, diagnosis/planning, preventive, restorative, endodontic, surgery/extraction, orthodontics, periodontics, oral rehabilitation) and prior dental anxiety history to address clinical heterogeneity.

Participant safety and ethics Participants may pause or stop the music or withdraw from the study at any time without impact on clinical care; any discomfort related to the use of headphones triggers immediate suspension of the intervention and clinical reassessment. Headphone volume is kept at a safe listening level to mitigate auditory risk, and all adverse events are recorded and managed per clinic policy. The study protocol has obtain ethics committee approval prior to enrollment, and all participants provide written informed consent; data are pseudonymized, stored on secure, access-restricted platforms, and managed to protect privacy and confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Adults receiving care at the university-affiliated dental clinic, legally able to consent and willing to participate voluntarily.
* Ability to read and independently complete brief self-report questionnaires before and after the visit.

Exclusion Criteria:

* Self-reported hearing impairment, current use of hearing aids, or other auditory conditions that interfere with safe headphone use or outcome validity.
* Use of sedative medication prior to the visit for the current appointment, or acute intoxication that may alter anxiety ratings.
* Cognitive impairment or other condition that limits capacity to provide informed consent or to complete study questionnaires reliably.
* Unwillingness to wear headphones during the procedure if randomized to a headphone arm, or refusal to participate/withdrawal of consent at any time.
* Any urgent clinical indication that, in the clinician's judgment, precludes headphone use (for example, need for uninterrupted verbal interaction or imaging incompatible with wearing the device).
* Reported history of severe adverse reactions to headphone use (for example, marked discomfort, vertigo) or skin sensitivity incompatible with device contact points.
* Inability to protect privacy or comply with basic study procedures (for example, cannot complete pre- and post-visit questionnaires within the clinic workflow)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
State Anxiety | Participants are assessed at the beginning and at the end of each dental appointment throughout a 5-month period
  State anxiety measured by the STAI Y-1 - State Anxiety Inventory
Dental anxiety | Participants are assessed at the beginning and at the end of each dental appointment throughout a 5-month period
  Dental anxiety measured by the MDAS - Modified Dental Anxiety Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Egas Moniz School of Health and Science, Almada, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zwiri A, Alam MK, Alshammari WA, Almazyad FM, Noor NFBM. Exploration of the Role of Music Therapy in Reducing Dental Anxiety. J Pharm Bioallied Sci. 2025 Jun;17(Suppl 2):S1273-S1275. doi: 10.4103/jpbs.jpbs_85_25. Epub 2025 Jun 18. PMID 40655808
- [Background] T Zaatar M, Alhakim K, Enayeh M, Tamer R. The transformative power of music: Insights into neuroplasticity, health, and disease. Brain Behav Immun Health. 2023 Dec 12;35:100716. doi: 10.1016/j.bbih.2023.100716. eCollection 2024 Feb. PMID 38178844
- [Background] Steenen SA, Linke F, van Westrhenen R, de Jongh A. Interventions to reduce adult state anxiety, dental trait anxiety, and dental phobia: A systematic review and meta-analyses of randomized controlled trials. J Anxiety Disord. 2024 Jul;105:102891. doi: 10.1016/j.janxdis.2024.102891. Epub 2024 Jun 24. PMID 38945067
- [Background] Shih KC, Hsu WT, Yang JL, Man KM, Chen KB, Lin WY. The Effect of Music Distraction on Dental Anxiety During Invasive Dental Procedures in Children and Adults: A Meta-Analysis. J Clin Med. 2024 Oct 29;13(21):6491. doi: 10.3390/jcm13216491. PMID 39518630
- [Background] Packyanathan JS, Lakshmanan R, Jayashri P. Effect of music therapy on anxiety levels on patient undergoing dental extractions. J Family Med Prim Care. 2019 Dec 10;8(12):3854-3860. doi: 10.4103/jfmpc.jfmpc_789_19. eCollection 2019 Dec. PMID 31879625
- [Background] Lee HY, Nam ES, Chai GJ, Kim DM. Benefits of Music Intervention on Anxiety, Pain, and Physiologic Response in Adults Undergoing Surgery: A Systematic Review and Meta-analysis. Asian Nurs Res (Korean Soc Nurs Sci). 2023 Aug;17(3):138-149. doi: 10.1016/j.anr.2023.05.002. Epub 2023 Jun 3. PMID 37276961
- [Background] Hao T, Pang J, Liu Q, Xin P. A systematic review and network meta-analysis of virtual reality, audiovisuals and music interventions for reducing dental anxiety related to tooth extraction. BMC Oral Health. 2023 Sep 22;23(1):684. doi: 10.1186/s12903-023-03407-y. PMID 37735362
- [Background] de Witte M, Pinho ADS, Stams GJ, Moonen X, Bos AER, van Hooren S. Music therapy for stress reduction: a systematic review and meta-analysis. Health Psychol Rev. 2022 Mar;16(1):134-159. doi: 10.1080/17437199.2020.1846580. Epub 2020 Nov 27. PMID 33176590
- [Background] Dalli OE, Yildirim Y, Aykar FS, Kahveci F. The effect of music on delirium, pain, sedation and anxiety in patients receiving mechanical ventilation in the intensive care unit. Intensive Crit Care Nurs. 2023 Apr;75:103348. doi: 10.1016/j.iccn.2022.103348. Epub 2022 Dec 2. PMID 36470699
- [Background] Crego A, Carrillo-Diaz M, Armfield JM, Romero M. From public mental health to community oral health: the impact of dental anxiety and fear on dental status. Front Public Health. 2014 Feb 28;2:16. doi: 10.3389/fpubh.2014.00016. eCollection 2014. PMID 24616889
- [Background] Aravena PC, Almonacid C, Mancilla MI. Effect of music at 432 Hz and 440 Hz on dental anxiety and salivary cortisol levels in patients undergoing tooth extraction: a randomized clinical trial. J Appl Oral Sci. 2020;28:e20190601. doi: 10.1590/1678-7757-2019-0601. Epub 2020 May 11. PMID 32401941
- [Background] Ainscough SL, Windsor L, Tahmassebi JF. A review of the effect of music on dental anxiety in children. Eur Arch Paediatr Dent. 2019 Feb;20(1):23-26. doi: 10.1007/s40368-018-0380-6. Epub 2018 Oct 29. PMID 30374854
- [Background] Aardal V, Willumsen T, Evensen KB. Differences in anxiety, depression, and oral health-related quality of life among dental anxiety patients with and without reported abuse experience. Eur J Oral Sci. 2024 Apr;132(2):e12976. doi: 10.1111/eos.12976. Epub 2024 Feb 2. PMID 38305706
- [Background] Aardal V, Evensen KB, Willumsen T, Hervik Bull V. The complexity of dental anxiety and its association with oral health-related quality of life: An exploratory study. Eur J Oral Sci. 2023 Feb;131(1):e12907. doi: 10.1111/eos.12907. Epub 2022 Nov 23. PMID 36418106